CLINICAL TRIAL: NCT05165719
Title: Validation of Specificity, Sensitivity, and Accuracy for an ELISpot-based In-vitro Diagnostic (IVD) Kit 'Corona-T-test' for Assessment of SARS-COV-2-specific T-cell Response
Brief Title: Validation of 'Corona-T-test' for Assessment of SARS-COV-2-specific T-cell Response After COVID-19 or Vaccination
Status: Completed | Type: Observational
Sponsor: National Research Center for Hematology, Russia (Network)
Collaborators: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other); DNKOM LLC (Other)
Responsible Party: Sponsor
Other Study IDs: Corona-T-test
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: SARS-CoV-2 Infection; SARS-CoV-2 Vaccination
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vaccinated: SARS-CoV-2 vaccination with 'Sputnik V' (Gam-COVID-Vac) in a period 7-14 days after the second vaccination before recruitment
  Interventions: Diagnostic Test: Corona-T-test
- Convalescents: PCR (polymerase chain reaction) confirmed COVID-19 in a period 14-45 days before recruitment
  Interventions: Diagnostic Test: Corona-T-test
- Healthy donors: No self-reported COVID-19 infection
  Interventions: Diagnostic Test: Corona-T-test

INTERVENTIONS:
Diagnostic Test: Corona-T-test — Corona-T-test - a single-color enzymatic ELISpot kit for the detection of interferon-gamma (IFNɣ), produced by the National Research Center for Hematology aiming detection of SARS-CoV-2-specific T cells

SUMMARY:
Accuracy validation of the designed and manufactured ELISpot-based in vitro diagnostic 'Corona-T-test' for detection of SARS-CoV-2-specific T cells.

DETAILED DESCRIPTION:
The investigators enrolled three independent cohorts of vaccinated (n = 69), convalescent (n = 50), and healthy but unvaccinated individuals (n = 101). Further, they estimated the T cell response to the designed peptide antigen panel, as measured by the manufactured ELISpot-based in vitro diagnostic 'Corona-T-test' to detect SARS-CoV-2-specific T cells.

ELIGIBILITY:
Non-specific inclusion criteria

* Participants aged 18 and above
* Participants agreeing to follow the study procedures
* Participants able to understand the purpose, nature, and methodology of the study
* Participants having signed the informed consent

Healthy donors inclusion criteria

* No self-reported COVID-19 infection
* No vaccination against COVID-19
* No immunoglobulin (Ig) IgM or IgG antibodies against SARS-CoV-2 by three tests (IgM to SARS-CoV-2 detection: "SARS-CoV-2-IgМ-ELISA-BEST", Ref #D-5502, IgG to SARS-CoV-2 S protein detection: "SARS-CoV-2-IgG-quantity-ELISA-BEST", "Vector-Best", Ref #D-5505), IgG to SARS-CoV-2 N protein detection: "SARS-CoV-2 IgG Reagent Kit", ARCHITECT, Abbott Laboratories, EU)

Convalescents inclusion criteria

* Self-reported COVID-19 infection
* PCR confirmed COVID-19 in a period 14-45 days before recruitment
* Detectable IgG antibodies against SARS-CoV-2 (IgG to RBD domain of SARS-CoV-2 S protein detection: "SARS-CoV-2-IgG-ELISA", "National Medical Research Center for Hematology", Moscow, Russia. Ref #K153G)

Vaccinated inclusion criteria

* SARS-CoV-2 vaccination with 'Sputnik V' (Gam-COVID-Vac) in a period 7-14 days after the second vaccination before recruitment
* Detectable IgG antibodies against SARS-CoV-2 (IgG to receptor-binding domain (RBD) domain of SARS-CoV-2 S protein: "SARS-CoV-2-IgG-ELISA", "National Medical Research Center for Hematology", Moscow, Russia. Ref #K153G)

Exclusion criteria

- Age under 18 y.o.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The attendees of the LTT 'DNKOM' were screened for the inclusion/exclusion criteria with a questionnaire and the above-mentioned serology tests.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
The result of Corona-T-test | 1 week
  positive, negative, or inconclusive (gray-zone)

CONTACTS AND LOCATIONS:
Overall Officials: Grigory A Efimov, MD PhD, Principal Investigator — National Research Center for Hematology
Locations (1):
- National Research Center for Hematology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No